CLINICAL TRIAL: NCT02935933
Title: Safety and Efficacy of Paravertebral Morphine Versus Dexmedetomidine on Acute and Chronic Pain
Brief Title: Paravertebral Morphine Versus Dexmedetomidine on Acute and Chronic Postmastectomy Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 347
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Acute Pain; Chronic Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Morphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paravertebral block with bupivacaine (Active Comparator): patients received 20 ml of bupivacaine 0.25% paravertebrally in 3 levels, divided into 6-7 ml in each level
  Interventions: Drug: bupivicaine
- Paravertebral block with bupivacaine + morphine (Active Comparator): patients received 20 ml of bupivacaine 0.25% +5 mg morphine paravertebrally in 3 levels, divided into 6-7 ml in each level.
  Interventions: Drug: bupivicaine; Drug: morphine
- Paravertebral block with bupivacaine + dexmedetomidine (Active Comparator): patients received 20 ml of bupivacaine 0.25% + 1 μg/kg dexmedetomidine paravertebrally in 3 levels divided into 6-7 ml in each level.
  Interventions: Drug: bupivicaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: bupivicaine — Paravertebral block
Drug: morphine
  Arms: Paravertebral block with bupivacaine + morphine
Drug: Dexmedetomidine
  Arms: Paravertebral block with bupivacaine + dexmedetomidine

SUMMARY:
Evaluate the effect of addition of morphine, dexmedetomidine to bupivacaine in PVB could improve the analgesic effect and thus reduce postoperative morphine consumption and development of chronic neuropathic pain, compared to PVB with bupivacaine , in patients undergoing major breast cancer surgery, i.e., modified radical mastectomy (MRM) and breast conservation surgery with axillary lymph node dissection.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed malignancy and a leading cause of cancer-related deaths among women. Surgery followed by chemotherapy and/or radiotherapy are the mainstay of current management. Chronic pain, or persistent postsurgical pain, which until recently was considered infrequent after breast cancer surgery (BCS), affects 60% to 80% of breast cancer survivors. The exact cause of chronic pain after BCS is not clear, but there is an association between acute postoperative pain and chronic pain generation after BCS. Postoperative pain intensity and analgesic consumption are significantly higher in patients who develop chronic pain after BCS, and it is suggested that optimizing postoperative pain management may reduce chronic pain. preoperative paravertebral block (PVB) administration in additional to general anesthesia, which has consistently been demonstrated to improve acute postoperative pain control and decrease length of hospital stay. The role of TPVB in preventing chronic pain is still evolving. Karmakar et al. shed more light on the impact of TPVBs in preventing and reducing the severity of chronic pain after breast surgery.

The discovery of peripheral opioid receptors led to the clinical application of adding opioids to local anesthetics for peripheral nerve blocks. Studies from the 1990s showed mixed results from the addition of morphine to peripheral nerve blocks, with two suggesting enhancement of analgesia duration and several showing no benefit at all.

Dexmedetomidine is a highly selective alpha-2 adrenoreceptor agonist that has been shown to have both sedative and analgesic effects. Although it is approved only for intravenous (IV) sedation, it has been extensively used for off-label indications, including neuraxial and peripheral nerve blocks, with good results. A significant prolongation of duration of analgesia has been reported when dexmedetomidine was added to LA for epidural analgesia, caudal block, subarachnoid block, PVB, brachial plexus block, ulnar nerve block and greater palatine nerve block.

ELIGIBILITY:
Inclusion Criteria:

* physical status classes I to III ( weight 50 - 85 kg), will be scheduled for unilateral modified radical mastectomy (MRM) with axillary evacuation will be consecutively enrolled.

Exclusion Criteria:

* patient refusal,
* patients with a known allergy to investigated drugs,
* bleeding disorders,
* anatomical abnormalities,
* infection in the paravertebral region,
* pregnancy, breast feeding,
* a history of drug or alcohol abuse, and patients with chronic pain or regularly receiving analgesics.
* patients subjected for bilateral mastectomy or any unilateral breast surgery other than MRM with axillary evacuation.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
total dose of morphine consumption | 48 hours
  the total dose of morphine consumption

SECONDARY OUTCOMES:
visual analouge scale | 0 (immediately after recovery from anesthesia), 2,4,6,12,24,36 and 48 hour postoperatively
  The pain intensity at rest (VAS-R) and arm movement of 90° (VAS-M) will be evaluated by VAS score at the same point of assessments.
chronic postmastectomy pain | 1,2,3 months
  The probability of developing chronic neuropathic pain will be assessed during regular postoperative examination in pain clinic in South Egypt Cancer Institute using LANSS ) in the 1st, 2nd and 3rd postoperative months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Iorg0006563, Egypt

IPD SHARING:
Plan to Share IPD: No